CLINICAL TRIAL: NCT01588145
Title: Phase I/II Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of HM61713 in NSCLC Patients With EGFR Mutation
Brief Title: Phase I/II Trial to Evaluate Safety, Tolerability and Pharmacokinetic Profile of HM61713 in NSCLC Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMSI-101
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; HM61713; EGFR-TKI; Phase II; olmutinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — olmutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM61713 (Experimental)
  Interventions: Drug: HM61713

INTERVENTIONS:
Drug: HM61713 — BID or QD, PO X 21 day cycle Number of cycles: until progression or unacceptable toxicity develops
  Other Names: Olmutinib

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of HM61713.

DETAILED DESCRIPTION:
Besides the main objective, there are 3 other objectives as follows:

* To evaluate the anti-cancer effect of HM61713 in NSCLC patients with EGFR mutation
* To investigate the pharmacokinetic profile of HM61713 and its metabolites after oral administration
* To investigate biomarkers related to the safety and efficacy of HM61713

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of advanced NSCLC
* Patients with EGFR mutation-positive tumor
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Estimated life expectancy of at least 12 weeks
* Subjects with adequate bone marrow (WBC ≥4,000/mm3, Platelet ≥100,000/mm3, Hemoglobin≥9.0g/dL, ANC≥1,500/mm3), renal (Creatinine≤1.5 mg/dl) and hepatic [aspartate aminotransferase (AST)/ alanine aminotransferase (ALT)/ alkaline phosphatase (ALP)≤3 x ULN, Total bilirubin ≤2.0 mg/dL] function. No significant heart and lung disease.

  ※ For subjects with a liver metastases, AST/ALT/ALP≤ 5 x ULN is allowed; and for subjects with bone marrow metastases, ALP≤ 5 x ULN is allowed
* Patients with amylase level ≤ 1.5 x ULN
* Subjects who have provided voluntary consent to participate in the study, and signed the written consent document

<Dose escalation part>

- Malignancy that has progressed after at least two prior chemotherapy regimens, including EGFR-TKI

<Expansion part 1>

* Patients with disease progression despite anticancer therapy with EGFR-TKI (e.g., erlotinib, gefitinib, neratinib, afatinib, dacomitinib)
* Patients who have provided voluntary consent for collection of tumor tissue taken and archived after the last anticancer therapy or collection of new tissue specimen and signed the written consent document

<Expansion part 2> & <Phase 2>

* Patients with disease progression despite anticancer therapy with EGFR TKI (e.g., erlotinib, gefitinib, neratinib, afatinib, dacomitinib) (Except treatment with EGFR mutation selective inhibitor, the same class of drug as investigational drug in this study)
* T790M mutation-positive confirmed in tissue collected after PD is confirmed during or after the last anticancer therapy
* At least one measurable target lesion allowing repeated measurement according to RECIST ver1.1 as of screening

<Phase 1 Expansion part 3>

* Patients with disease progression despite anticancer therapy with EGFR TKI (e.g., erlotinib, gefitinib, neratinib, afatinib, dacomitinib) (Except treatment with EGFR mutation selective inhibitor, the same class of drug as investigational drug in this study)
* T790M mutation-negative confirmed in tissue collected after progressive disease (PD) is confirmed during or after the last anticancer therapy
* At least one measurable target lesion allowing repeated measurement according to RECIST ver1.1 as of screening

Exclusion Criteria:

* Hematologic malignancies
* Symptomatic or uncontrolled central nervous system metastases
* Interstitial lung disease, including pulmonary fibrosis
* LVEF < 40% or NYHA Class III or IV heart failure
* History of pancreatitis
* History or current evidence, of any psychiatric or congenital disorder, including dementia or epilepsy
* Compromised organ function, infection or allergy
* Pregnant or breast-feeding women, or women of child-bearing potential who do not use an appropriate method of contraception (male patients should also use an appropriate method of contraception during the study period)
* Patients who had received other investigational product within 30 days prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2012-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Dose limiting Toxicity will be evaluated on Day 24 during Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wan Kim, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul, South Korea